CLINICAL TRIAL: NCT01983319
Title: Transcranial Direct Current Stimulation Combined With Constraint Induced Movement Therapy and Role of GABA Activity in Stroke Recovery
Brief Title: tDCS Combined With Constraint Induced Movement Therapy and Role of GABA Activity in Stroke Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Regionshospitalet Hammel Neurocenter (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Krystian Figlewski, MD, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M-2013-268-13
Record Dates: First submitted 2013-10-31; First posted 2013-11-13 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation; Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- CIMT + active anodal tDCS (Experimental): Subjects in this group will be trained with constraint-induced movement therapy for the hand (10 consecutive sessions Monday- Friday) while concurrently receiving active anodal transcranial Direct Current Stimulation 1,5 mA for 30 min.
  Interventions: Device: active anodal transcranial Direct Current Stimulation (tDCS); Behavioral: Constraint Induced Movement Therapy (CIMT)
- CIMT + sham tDCS (Sham Comparator): Subjects in this group will be trained with constraint-induced movement therapy for the hand (10 consecutive sessions Monday- Friday) while concurrently receiving sham transcranial Direct Current Stimulation
  Interventions: Device: sham transcranial Direct Current Stimulation; Behavioral: Constraint Induced Movement Therapy (CIMT)
- Healthy control subjects (No Intervention): 20 healthy age-matched control subjects will undergo MRI spectroscopy of the brain.

INTERVENTIONS:
Device: active anodal transcranial Direct Current Stimulation (tDCS) — Anodal transcranial Direct Current Stimulation 1.5 mA in 30 minutes with CIMT
  Other Names: tDCS; Non invasive brain stimulation; transcranial stimulation
  Arms: CIMT + active anodal tDCS
Device: sham transcranial Direct Current Stimulation — sham transcranial Direct Current Stimulation 30 min with CIMT
  Other Names: placebo stimulation
  Arms: CIMT + sham tDCS
Behavioral: Constraint Induced Movement Therapy (CIMT) — 2 weeks of CIMT
  Other Names: CIMT
  Arms: CIMT + active anodal tDCS; CIMT + sham tDCS

SUMMARY:
The aim of this study is to determine whether noninvasive brain stimulation in form of active transcranial direct current stimulation (tDCS) combined with constraint induced movement therapy (CIMT) offers an additional benefit as compared with sham tDCS combined with CIMT in patients with stroke. Furthermore the purpose is to highlight changes in GABA activity more than 3 months after stroke and its importance for effect of tDCS and CIMT combined with tDCS.

ELIGIBILITY:
Inclusion Criteria:

* stroke onset >3 months prior to study enrollment
* subject has at least 10 degrees mobility over wrist, thumb and fingers on the affected side
* subject can move, stand up and stand firmly with constrained healthy hand
* subject can perform training 6 hours daily in 2 weeks
* subject is able to understand instructions and be able to cooperate

Exclusion Criteria:

* pregnancy
* contraindications to MRI of brain
* epilepsy, major psychiatric disease
* excessive pain that prevents training
* history of other diseases resulting decreased mobility of affected upper limb

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in Upper Limb function | Baseline and posttest (an average of 2 weeks from baseline)
  The motor function assessment will be done with: Wolf Motor Function Test

SECONDARY OUTCOMES:
GABA (gamma-aminobutyric acid) activity | Baseline
  Assessment of GABA activity using MRI spectroscopy. Measurements will be compared between patients undergoing CIMT and healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Henning Andersen, Professor, Study Director — Aarhus University Hospital
Locations (1):
- Regionhospital Hammel Neurocenter, Research Unit, Hammel, Denmark

REFERENCES:
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411
- [Derived] Figlewski K, Blicher JU, Mortensen J, Severinsen KE, Nielsen JF, Andersen H. Transcranial Direct Current Stimulation Potentiates Improvements in Functional Ability in Patients With Chronic Stroke Receiving Constraint-Induced Movement Therapy. Stroke. 2017 Jan;48(1):229-232. doi: 10.1161/STROKEAHA.116.014988. Epub 2016 Nov 29. PMID 27899754